CLINICAL TRIAL: NCT07304518
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging Phase II Trial of PRT-064040 Nasal Spray for the Acute Treatment of Migraine
Brief Title: Phase II Trial of PRT-064040 Nasal Spray for the Treatment of Migraine in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Purity Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-PRT-064-201
Record Dates: First submitted 2025-12-03; First posted 2025-12-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PRT-064040 nasal spray (dose 1) (Experimental): Participants administered a single intranasal dose of PRT-064040 nasal spray (dose 1) on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization.
  Interventions: Drug: PRT-064040 nasal spray
- PRT-064040 nasal spray (dose 2) (Experimental): Participants administered a single intranasal dose of PRT-064040 nasal spray (dose 2) on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization.
  Interventions: Drug: PRT-064040 nasal spray
- PRT-064040 nasal spray (dose 3) (Experimental): Participants administered a single intranasal dose of PRT-064040 nasal spray (dose 3) on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization.
  Interventions: Drug: PRT-064040 nasal spray
- Placebo (Experimental): Participants administered a single intranasal dose of placebo on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRT-064040 nasal spray — A single dose of PRT-064040 nasal spray
  Arms: PRT-064040 nasal spray (dose 1); PRT-064040 nasal spray (dose 2); PRT-064040 nasal spray (dose 3)
Drug: Placebo — A single dose of placebo matched to PRT-064040 nasal spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about the efficacy and safety of PRT-064040 Nasal Spray versus placebo in the acute treatment of moderate or severe migraine.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

1. Male and female participants aged 18-75 years (inclusive);
2. BMI < 35 kg/m²;
3. Participant has at least 1-year history of migraines (with or without aura), consistent with a diagnosis according to the International Classification of Headache Disorder, 3rd Edition;
4. Age at first migraine onset < 50 years;
5. Migraine attacks, on average, lasting about 4-72 hours if untreated or treatment-resistant;
6. 2-8 attacks of moderate to severe intensity per month within the last 3 months；
7. Less than 15 days with headache (migraine or non-migraine) per month within the last 3 months；
8. Participants on prophylactic migraine medication are permitted to remain on therapy provided they have been on a stable dose for at least 3 months prior to screening visit and the dose is not expected to change until the EOT visit;
9. Patients diagnosed with chronic migraine who, owing to stable preventive therapy, have < 15 headache days and 2-8 attacks of moderate to severe intensity per month in the 3 months before screening, and who meet all other entry criteria, may be enrolled;
10. Able to comprehend and complete study questionnaires with electronic patient-reported outcome (e-PRO) application.

Exclusion Criteria:

Key Exclusion Criteria:

1. Participant with history of migraine with brainstem aura, retinal migraine, or hemiplegic migraine.
2. Participant with evidence of poorly controlled, unstable, or recently diagnosed cardiovascular or cardiometabolic disease, or prior history thereof, including:

   * Ischemic heart disease, coronary vasospasm, or cerebral ischemia diagnosed within 6 months before screening;
   * Previous stroke, transient ischemic attack, myocardial infarction, acute coronary syndrome, cardiac surgery, or percutaneous coronary intervention;
   * Abnormal 12-lead ECG at screening;
   * Poorly controlled diabetes mellitus or hypertension;
   * Poorly controlled or severe peripheral vascular disease.
3. Participant with any nasal structural abnormality, mucosal lesion, or disorder that could interfere with intranasal drug absorption.
4. Participant with dysgeusia, hypogeusia, or related taste disorders.
5. Participant with acute or chronic pain syndromes, or any other pain that in the investigator's opinion could confound study assessments.
6. Participant with history of regular use of ergotamine or triptans ≥ 10 days per month for ≥ 3 months; or regular use of non-narcotic analgesics (e.g., acetaminophen, NSAIDs, gabapentin) ≥ 15 days per month for ≥ 3 months.
7. Clinically relevant abnormal findings in hepatitis B surface antigen, hepatitis C antibody, Treponema pallidum antibody, or HIV antibody tests at screening.
8. Participant with history of alcohol or drug abuse within 1 year before screening, or positive urine drug screen at screening.
9. Pregnant or lactating women, or positive pregnancy test at screening.
10. Participant with known hypersensitivity to the investigational product or any of its excipients, or history of significant allergic reactions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Freedom From Pain at 2 Hours Post-dose | 2 hours post-dose
Percentage of Participants With Freedom From Most Bothersome Symptom (MBS) at 2 Hours Post-dose | 2 hours post-dose

SECONDARY OUTCOMES:
Percentage of Participants With Pain Relief at 15 Minutes Post-dose | 15 minutes post-dose
Percentage of Participants With Pain Relief at 30 Minutes Post-dose | 30 minutes post-dose
Percentage of Participants With Pain Relief at 60 Minutes Post-dose | 60 minutes post-dose
Percentage of Participants With Pain Relief at 2 Hours Post-dose | 2 hours post-dose
Percentage of Participants Who Were Able to Function Normally at 2 Hours Post-dose | 2 hours post-dose
Percentage of Participants With Sustained Pain Relief From 2 Hours to 24 Post-dose | From 2 to 24 hours post-dose
Percentage of Participants With Sustained Pain Relief From 2 Hours to 48 Post-dose | From 2 to 48 hours post-dose
Percentage of Participants Who Were Able to Function Normally at 30 Minutes Post-dose | 30 minutes post-dose
Percentage of Participants Who Were Able to Function Normally at 60 Minutes Post-dose | 60 minutes post-dose
Percentage of Participants With Freedom From Phonophobia at 2 Hours Post-dose | 2 hours post-dose
Percentage of Participants With Freedom From Photophobia at 2 Hours Post-dose | 2 hours post-dose
Percentage of Participants With Freedom From Nausea at 2 Hours Post-dose | 2 hours post-dose
Percentage of Participants With Sustained Pain Freedom From 2 Hours to 24 Post-dose | From 2 to 24 hours post-dose
Percentage of Participants With Sustained Pain Freedom From 2 Hours to 48 Post-dose | From 2 to 48 hours post-dose
Percentage of Participants With Pain Relapse From 2 to 48 Hours Post-dose | From 2 hours to 48 hours post-dose
Percentage of Participants With Rescue Medication Use Within 24 Hours Post-dose | Through 24 hours post-dose
Percentage of Participants Who Were Able to Function Normally at 15 Minutes Post-dose | 15 minutes post-dose
The incidence and severity of adverse events | Through 7(±2) days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- The First Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No